CLINICAL TRIAL: NCT03366142
Title: Use of Ustekinumab (Anti-IL-12/23p40 Monoclonal Antibody) in Patients With Leukocyte Adhesion Deficiency Type 1 (LAD1) Who Have Inflammatory Pathology
Brief Title: Ustekinumab (Anti-IL-12/23p40 Monoclonal Antibody) in Patients With Leukocyte Adhesion Deficiency Type 1 (LAD1) Who Have Inflammatory Pathology
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180022; 18-I-0022
Record Dates: First submitted 2017-12-07; First posted 2017-12-08 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10-18

CONDITIONS: LAD1
Keywords: Autosomal Recessive Disorder; Immune; Gingival; Oral Ulcer; Cytokine Expression
MeSH Terms: conditions — Oral Ulcer | interventions — Ustekinumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): treatment with ustekinumab based on weight
  Interventions: Drug: Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab — 0.75 mg/kg or 45 or 90 mg via subcutaneous injection for 5 doses (second dose 4 weeks after first, subsequent doses every 12 weeks thereafter).

SUMMARY:
Background:

The disease leukocyte adhesion deficiency type 1 (LAD1) affects white blood cells. Those are immune system cells. In people with LAD1, white blood cells do not properly communicate with the rest of the body. This causes uncontrolled inflammation, particularly in the gums. People with LAD1 can get frequent infections and tend to lose their teeth before adulthood. Researchers want to see if a drug called ustekinumab helps people with LAD1.

Objective:

To study the safety and tolerability of ustekinumab in treating gum inflammation in people with LAD1.

Eligibility:

People ages 12 65 with LAD1

Design:

Participants will be screened with:

* Medical history
* Physical exam
* Oral exam
* A scan of the chest, abdomen, and pelvis for possible infection
* Blood and urine tests

The baseline visit will take 2 days. Participants will:

* Repeat most screening tests
* Have a skin exam
* Have small pieces of their gums removed (biopsy)
* Have mouth fluids collected
* Get the study drug injected under the skin of the abdomen, thigh, or elsewhere on the body. They will be watched for at least 2 hours.

Participants will be instructed on tracking how they are feeling and any side effects.

Participants will have 4 more visits over 40 weeks. They will get the study drug and repeat the baseline tests.

Participants may have up to 5 more tissue biopsies.

Participants will be called between visits to discuss how they are feeling and side effects.

Participants will have a final visit 52 weeks after the baseline. They will repeat most of the baseline tests.

Participants will answer questions about their oral ulcers.

DETAILED DESCRIPTION:
Lymphocyte adhesion deficiency type 1 (LAD1) is an autosomal recessive disorder of leukocyte function. Decreased expression of the <=2 subunit of leukocyte integrins results in abnormal cell-cell and cell extracellular matrix adhesion. This disease is characterized by recurrent bacterial infections, impaired wound formation, and other aberrations of adhesion-dependent functions. The severe phenotype can be fatal, but patients with even moderate phenotypes are prone to infection and lose their teeth despite treatment.

Ustekinumab is a monoclonal antibody directed against the p40 subunit of human interleukins IL-12 and IL-23. It is approved for treatment of moderate-to-severe plaque psoriasis, active psoriatic arthritis, and moderate-to-severe Crohn s disease. By binding the shared p40 subunit of IL-12 and IL-23, ustekinumab exerts clinical effects through interruption of the TH1 and TH17 cytokine pathways. Previous work at the NIH suggests that blockade of IL-17, which is highly expressed in the gingiva of people with LAD1, can reduce bacterial load and resolve inflammatory gingival disease. We have treated one patient with ustekinumab for 1 year; during this time, he had no serious infections and there was a dramatic resolution of his inflammatory lesions. Our goal is to explore the potential of ustekinumab as treatment for LAD1 inflammatory disease.

The objective of this open-label, proof-of-concept study is to evaluate the safety and tolerability of ustekinumab in 10 patients with LAD1. Participants will receive 5 doses of ustekinumab via subcutaneous injection over the course of 1 year. They will be evaluated for adverse events, as well as the effect of the drug on inflammatory lesions and biomarker expression.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 12-65 years.
* Molecularly and cellularly confirmed LAD1 with inflammatory lesions.
* Willing to allow storage of biological samples for future research.
* Willing to allow genetic testing of blood samples.
* Able to provide informed consent.
* Participants who can get pregnant or impregnate a partner must agree to use adequate contraception when engaging in sexual activities that can result in pregnancy. Adequate contraception must be used consistently starting at screening and lasting through the final study visit. Appropriate forms of contraception include the following:

  1. Intrauterine device or equivalent.
  2. Hormonal contraceptive (eg, consistent, timely, and continuous use of contraceptive pill, patch, ring, implant, or injection) that has reached full efficacy before dosing.
  3. A double barrier method (eg, male/female condom, cap, or diaphragm plus spermicide).
  4. Be in a stable, long-term monogamous relationship, per assessment of the principal investigator (PI), with a partner who does not pose any potential pregnancy risk, eg, has undergone a vasectomy at least 6 months before the first dose of study agent or is of the same sex as the participant.
  5. Have had a hysterectomy and/or a bilateral tubal ligation or both ovaries removed.

EXCLUSION CRITERIA:

* History of malignancy (except for basal cell carcinoma) within the previous 5 years.
* Infected with HIV.
* Active uncontrolled bacterial, viral, or fungal infection.
* Active or chronic viral hepatitis.
* Active or latent untreated tuberculosis.
* Received Bacillus Calmette-Guerin vaccine within the last year.
* Received live attenuated vaccines within 15 weeks before the first dose.
* Allergy to any component of the ustekinumab formulation.
* Pregnant or breastfeeding.
* Any condition that, in the opinion of the investigator, contraindicates participation in this study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-07-02 (Actual); Primary Completion 2024-10-16 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of ustekinumab in treating LAD1 affected patients who have inflammation, such as gingival, skin or gut. | 13 months
  alteration of local gingival cytokine expression and peripheral blood cytokine expression, assessment of oral inflammation via gingival bleeding on probing measurements and changes to oral ulcer, lesions or gastro-intestinal inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz E Marciano, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share human data generated in this study for future research as follows:@@@-Identified data in the Biomedical Translational Research Information System (BTRIS, automatic for activities in the NIH CC).@@@-De-identified or identified data with approved outside collaborators under appropriate agreements.@@@-Data sharing may be complicated or limited in certain cases by contractual obligations or agreements with outside collaborators, such as cooperative research and development agreements, clinical trial agreements, other restraints, etc.
Supporting Information: SAP
Time Frame: @@@@@@IPD will become available after completion of the study@@@@@@Since LAD1 is a rare immune deficiency, we may reevaluate when IPD and associated sharing plan will be available as we approach the sample size.
Access Criteria: Data will be shared through:@@@-BTRIS (automatic for activities in the NIH CC).@@@-Approved outside collaborators under appropriate individual agreements.@@@-Publication and/or public presentations.@@@Data might be shared before publication.@@@The PI and MAI will review and approve requests.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2018-I-0022.html